CLINICAL TRIAL: NCT04387695
Title: SBRT Sequential TACE Combined With Sorafenib Versus Sorafenib Alone in the Treatment of Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus：A Single-center Randomized Controlled Study
Brief Title: SBRT+TACE+Sorafenib Vs Sorafenib in the Treatment of uHCC With PVTT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPIC2001
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Unresectable Hepatocellular Carcinoma; Portal Vein Thrombosis
Keywords: Hepatocellular Carcinoma,Portal Vein Tumor Thrombus; Radiation ,Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT + TACE + Sorafenib (Experimental): SBRT sequential TACE combined with Sorafenib
  Interventions: Radiation: SBRT+TACE+Sorafenib
- Sorafenib (Active Comparator): Sorafenib 800 mg/day orally
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Radiation: SBRT+TACE+Sorafenib — SBRT first for the PVTT +TACE for HCC within a week next +Sorafenib with 2 weeks later
  Other Names: Stereotactic Body Radiation Therapy
  Arms: SBRT + TACE + Sorafenib
Drug: Sorafenib — Sorafenib 800 mg/day orally
  Other Names: Nexavar
  Arms: Sorafenib

SUMMARY:
To evaluate and compare the efficacy and safety of SBRT sequential TACE combined with sorafenib versus sorafenib alone in the treatment of unreactable HCC with PVTT.

DETAILED DESCRIPTION:
HCC Patients classified as BCLC stage C present with PVTT, and the recommended first-line treatment is systemic therapy with sorafenib according to updated Barcelona Clinical Liver cancer (BCLC) treatment algorithms.However, recent data from observational studies suggest that the combination of TACE and SBRT would be as effective as sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Child-Pugh score ≤ 7
* Performance status: ECOG score ≤ 2
* HCC diagnosed by biopsy or by the noninvasive criteria of the Chinese Liver Cancer Guideline 2017
* the primary HCC being unresectable (BCLC C stage/ CNLC Ⅲa-b) according to NCCN guideline
* No previous therapy for HCC
* at least one measurable target lesion according to RECIST 1.1
* Adequate hematopoietic function: Hemoglobin ≥ 8.5 g/dL; Absolute neutrophil count ≥ 750/mm3; Platelet count ≥ 50,000/mm3
* Serum total bilirubin ≤ 2 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase ≤ 10 x ULN
* Creatinine ≤ 1.5 x ULN
* No plan for pregnancy or breast feeding. Active contraception.
* Willing to give informed consent

Exclusion Criteria:

* Prior history to or exposure of transarterial chemoembolization, external beam radiation to liver, or sorafenib
* Complete obstruction of hepatic outflow
* Uncontrolled ascites of hepatic encephalopathy
* Prior liver transplantation
* Positive for human immunodeficiency virus (HIV)
* Active gastric or duodenal ulcer
* Other uncontrolled comorbidities or malignancy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | at 12 weeks after randomization
  Progression is defined as progressive disease (PD) by independent radiologic review according to mRECIST criteria, termination of the assigned treatment, or death from any cause, assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons with the intention-to-treat principle.

SECONDARY OUTCOMES:
Radiologic response rate | at 12 weeks after randomization
  Radiologic response rate by independent radiologic review according to mRECIST criteria , assessed by Chi-square test or Fisher's exact test, as appropriate.
Overall patient survival rate | up to 2 years after randomization
  The median overall patient survival rate assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons.
Objective response rate | at 12 weeks and up to 2 years after randomization
  Objective response rate by independent radiologic review according to mRECIST criteria , assessed by Chi-square test or Fisher's exact test, as appropriate.
Disease control rate | at 12 weeks and up to 2 years after randomization
  Disease control rate by independent radiologic review according to mRECIST criteria , assessed by Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-hui Sun, MD,PH.D, Study Director — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No